CLINICAL TRIAL: NCT04282772
Title: Ectopic Eruption of Permanent First Molars: A Retrospective Study
Brief Title: Ectopic Eruption of Permanent First Molars
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Seçil Çalışkan, Assistant Professor, Eskisehir Osmangazi University
Other Study IDs: 2019/77-12
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Failure of Tooth Eruption Associated With Tooth Impaction
Keywords: Ectopic Eruption; Eruption Failure; Impacted Teeth
MeSH Terms: conditions — Tooth, Unerupted; Tooth, Impacted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ectopic Eruption: The ectopic eruption of PFMs were classified in two ways: impacted and self-corrected.
  Interventions: Diagnostic Test: Impacted; Diagnostic Test: Self-corrected

INTERVENTIONS:
Diagnostic Test: Impacted — Until an active treatment for the PFM is started or the early exfoliation of PSM occurs, the tooth remains in a self-locking position
Diagnostic Test: Self-corrected — The ectopic erupted permanent molar can disregard the self-locking position and continue in a normal direction, but the distal root of the PSM remains more or less a significant atypical resorption

SUMMARY:
Ectopic eruption may be defined as the eruption of a permanent tooth that takes place in such a manner that a partial or a total resorption of the root(s) of an adjacent primary tooth occurs and can be noted during routine dental radiographic evaluation. It is a common case in mixed dentition and is usually diagnosed by a pediatric dentist. This retrospective study aimed to determine the prevalence and related factors of the ectopic eruption of permanent first molars(PFM). This retrospective study was performed using the panoramic radiographs of 11,924 child patients aged 6-10 years with at least one ectopically erupted PFM were included. The total prevalence of ectopic eruption, type, age, gender, jaw distribution, and bilateral versus unilateral occurrence were determined. The angulation of PFM, mesialization ratio of PFM, and degree of adjacent primary second molar(PSM) tooth root resorption were also assessed. The chi-square test, ANOVA was used for statistical analysis. A total of 76 ectopic eruptions were detected in the maxilla, 6 in the mandible, and 2 in both the maxilla and the mandible. In terms of the eruption status of cases with ectopic eruption, 27 were self-corrected, 51 remained impacted, and 6 were both. The impaction rate of the right upper PFMs was higher than that of others. No significant relationship was found between eruption status and degree of resorption. As a conclusion, small impaction of the PFM does not mean that the PSM lesion is also small. With substantial displacements, a proportionally diminutive lesion can exist, and vice versa.

DETAILED DESCRIPTION:
Assessment of Angulation The angles between the axes of the PSMs and the long axes of the PFMs were measured. The angle was measured using ImageJ application (1.50 n, National Institutes of Health, Bethesda, MD, USA). The long axes were formed by a line extending parallel to the center of the tooth in an occluso-cervical manner. The vertical angle was defined as (-) or (+) according to Sun et al.The angles between the occlusal lines of the PSMs and the PFMs were measured. The horizontal angle was defined as (-) or (+) according to Sun et al.

Assessment of PSM Root Resorption The distal root resorption level of the PSM was determined using Barberia-Leache et al.'s classification2 as follows; Grade I: mild-limited resorption of the cementum or with minimum dentin penetration Grade II: moderate-resorption of the dentin without pulp exposition Grade III: severe-resorption of the distal root leading to pulp exposure Grade IV: very severe-resorption that affects the mesial root of the PSM.

Assessment of PFM Mesialization Ratio The mesiodistal size of the PFM and the amount of mesialization were measured by the Image J application to evaluate the differences between reversible and irreversible ectopic eruption. The mesiodistal size was measured from the largest part of the crown, and the amount of mesialization was measured using the distance between the drawn tangent on the distal wall of the PSM and the mesial convexity of the PFM. Afterwards, the amount of mesialization was proportioned to the mesiodistal size of the PFM.

ELIGIBILITY:
Inclusion Criteria:

-Among the 11,924 radiographs, only the children who had at least one ectopically erupted PFM were included.

Exclusion Criteria:

-Presence of any history of extraction due to impaction, orthodontic treatment, or caries; the presence of any craniofacial anomalies, congenital deformities, or syndromes involving dental eruption; absent adjacent PSMs; and presence of any cyst, tumor, or other pathological condition in the molar area.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 11,924 child patients aged 6-10 years who attended the Pediatric Dentistry clinics at the Faculty of Dentistry, Eskisehir Osmangazi University, between March 2016 and March 2018.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Determination of the ectopic eruption prevalence. | 6 months
  Data were collected retrospectively from clinical notes and panoramic radiographs. Among the 11,924 radiographs, only the children who had at least one ectopically erupted PFM were included.
Determination of the ectopic eruption related factors. | 3 months
  The angulation of PFM, mesialization ratio of PFM, and degree of adjacent PSM tooth root resorption were assessed using ImageJ application.

CONTACTS AND LOCATIONS:
Overall Officials: Seçil Çalışkan, Principal Investigator — Eskişehir Osmangazi University
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided